CLINICAL TRIAL: NCT06007469
Title: Pedal Acceleration Time (PAT) Versus Toe Brachial Pressure Index (TBPI) as a Measure of Foot Perfusion - A Pilot Study.
Brief Title: Pedal Acceleration Time (PAT) as a Measure of Foot Perfusion
Acronym: PAT
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Liverpool University Hospitals NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: SP0721
Record Dates: First submitted 2022-05-27; First posted 2023-08-23 (Actual); Last update posted 2023-08-23 (Actual); Status verified 2023-08

CONDITIONS: Critical Limb Ischemia; Claudication, Intermittent
Keywords: ischaemia; ABPI; TBPI; claudication; ulceration; acceleration time; duplex ultrasound
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia; Intermittent Claudication; Ischemia; Ulcer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Critical Limb Threatening Ischaemia: Patients presenting with Critical Limb Threatening Ischaemia
- Non-limb threatening peripheral vascular disease: Patients presenting with non-limb threatening peripheral vascular disease

SUMMARY:
To identify a correlation between Toe Brachial pressure Index (TBPI) and Acceleration time of the pedal vessels. The aim would then to use this data to design a clinical study assessing the relationship between PAT and wound healing in patients with PAD.

DETAILED DESCRIPTION:
The use of ankle brachial pressure index (ABPI) is commonplace in the screening, diagnosis and management of peripheral vascular disease (PAD). This technique measures and compares the occlusion pressure of the brachial arteries for comparison with the occlusion pressure of the tibial arteries at the level of the ankle. The index is then calculated by dividing the highest of the tibial occlusion pressures by the highest brachial occlusion pressure. In normal subjects the ABPI should fall between 09-1.3 (1) . A pressure less than 0.9 suggest a compromise to the peripheral circulation (PAD), with the blood pressure at the ankle level being lower than in the arm. ABPI results can be erroneous in the presence of medial artery calcification (MAC) where the ankle arteries are more difficult to compress and hence give falsely elevated readings. In some patients it can be impossible to occlude the arterial flow as the vessel is so rigid (1). Conditions that increase the prevalence of MAC are diabetes mellitus, chronic kidney disease as well as advancing age which also increased the stiffness of the vessel walls having a similar effect as MAC (2).

When used in isolation as a PAD screening, ABPI can give a normal reading due to undiagnosed pathological vessel stiffness with studies reporting up to 14-27% of patients returning normal ABPI results at the same time as low TBPI. (3) Despite the potential pitfall of ABPI, it is still a widely recognized as its diagnostic limits have been validated in several large scale studies. (3) However, due to the level of arterial assessment, ABPI does not actually assess circulation into the foot itself (4). The toe vessels are much less susceptible to vessel stiffness (3) , and hence deemed are more reliable in such cases when the ABPI would return a falsely elevated result.

When used alongside detailed duplex imaging of the peripheral arterial tree to give image guided documentation of vessel calcification, TBPI is a useful indicator of perfusion into the foot when the ABPI is known not to be indicated. Therefore TBPI measurement has become the established method for assessing arterial perfusion to the foot, particularly in patients with risk factors for MAC.

When investigating perfusion into the critically ischaemic limb, ABPI is not indicated and therefore TBPI is the preferred method. However this becomes problematic when there has been previous amputation of the forefoot/toes, the patient is in significant pain and/or there is tissue loss which impedes accurate placement of the equipment on the affected limb. Furthermore, in a significant number of these patients it is not possible to obtain an adequate waveform in the toe due to poor arterial perfusion.

To overcome this predicament a novel technique has been developed which involves direct ultrasound imaging of the pedal vasculature and use the systolic rise time calculated from the returned waveform analysis as a surrogate for ABPI (4) This systolic rise time, known as pedal acceleration time (PAT) in foot vessels, has been has been reported to correlate well with ABPI in patients with compressible vessels and therefore is felt to be a predictor of wound healing following direct and indirect revascularization. (4) There are, however, a significant group of patients that attend the vascular department that have risk factors for MAC which make them unsuitable for ABPI. For this group of patients and those with coexisting with foot wounds/previous amputation, there is no ratified method for investigation perfusion pressure.

The aim of this pilot study is to gather information from all patients who present with significant PAD to investigate a possible link between PAT, ABPI and TBPI and if PAT is a reliable measurement in patients who fall outside of the group normally excluded.

This would allow objective perfusion information and therefore guide treatment and management plans.

ELIGIBILITY:
Inclusion Criteria:

* 1. Male/Female 2. Adults aged 18 and above 3. Willing to provide written, informed consent 4. Referred into the vascular service with symptoms or confirmed PVD/CLTI

Exclusion Criteria:

1. Referral not indicative of PVD
2. Occlusion of vessels/no visible flow at the site of interest
3. Amputation of the limb
4. Tissue loss preventing assessment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients will be identified who attend the vascular clinic at the Royal Liverpool Hospital. The first 30 patients with critical limb threatening ischaemia (CLTI) that are identified and consent for the study will be recruited. Similarly the first 20 patients who have symptoms suggestive of non-critical, peripheral arterial disease such as intermittent claudication will be recruited.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-10-04 (Estimated); Primary Completion 2023-12-10 (Estimated); Study Completion 2024-12-03 (Estimated)

PRIMARY OUTCOMES:
Foot Perfusion. | 1 measure
  ankle arterial acceleration time versus toe pressure (mmHg) Manual blood pressures of at the toe (mmHg) will also be measured from all participants, where technically possible.